CLINICAL TRIAL: NCT03669601
Title: A Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of Ascending Doses of Combined Therapy With ATR Inhibitor AZD6738 and Gemcitabine, Using a Model Based Design.
Brief Title: AZD6738 & Gemcitabine as Combination Therapy
Acronym: ATRiUM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Professor Duncan Jodrell, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATRiUM
Record Dates: First submitted 2018-08-07; First posted 2018-09-13 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Cancer
Keywords: solid tumour; locally advanced; metastatic
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — ceralasertib; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Continuous and intermittent administration schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous AZD6738 & gemcitabine (Experimental): Intravenous gemcitabine on days 3, 10 and 17 of a 28 day cycle. Dose range from 500mg/m2 to 1000mg/m2.
  Oral tablet AZD6738 once daily for 21 days of a 28 day cycle. Dose range from 40mg to 120mg.
  Interventions: Drug: AZD6738; Drug: Gemcitabine
- Intermittent AZD6738 & gemcitabine (Experimental): Intravenous gemcitabine on days 3, 10 and 17 of a 28 day cycle. Dose range from 500mg/m2 to 1000mg/m2.
  Oral tablet AZD6738 once daily and intermittently for up to 12 days of a 28 day cycle. Dose range from 40mg to 120mg.
  Interventions: Drug: AZD6738; Drug: Gemcitabine

INTERVENTIONS:
Drug: AZD6738 — A potent, selective inhibitor of the serine/threonine-specific protein kinase, ataxia telangiectasia and Rad3-related protein (ATR), with good selectivity against other phosphatidylinositol 3-kinase-related kinase (PIKK) family members.
Drug: Gemcitabine — Nucleoside metabolic inhibitor.
  Other Names: Gemzar

SUMMARY:
A dose escalation trial to assess the safety of AZD6738 in combination with gemcitabine in participants with advanced solid tumours.

DETAILED DESCRIPTION:
A phase 1, non-randomised, multicentre, model-based dose escalation trial. This trial will assess the safety, tolerability, pharmacokinetics and preliminary anti-tumour activity of ascending doses of combined therapy with ATR inhibitor (AZD6738) and gemcitabine, in participants with advanced solid tumours, followed by an expansion phase in participants with advanced pancreatic ductal adenocarcinoma (PDAC).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate.
* Aged 18 years and over.
* ECOG performance status of 0 or 1.
* Dose escalation phase only: Patients with inoperable/unresectable, histologically proven, locally advanced or metastatic solid tumour that has progressed on standard therapy, or patients unwilling to receive standard therapy.
* Treatment expansion phase only: Patients with inoperable, histologically proven, locally advanced or metastatic pancreatic adenocarcinoma that has progressed on conventional chemotherapy, or patients unwilling to receive standard therapy.
* Documented evidence of progression (radiological or clinical) prior to trial entry.
* Estimated life expectancy of ≥12 weeks.
* Measurable tumour lesions that can be accurately assessed at baseline by computed tomography (CT) and are suitable for repeated assessment as per RECIST 1.1 and considered accessible for core biopsy.
* Women of childbearing potential, male participants and their partners are required, and must be willing, to use 2 highly effective forms of contraception for the duration of the trial and for six (6) months after the completion of the trial treatment (see section 11.13). Women of non-childbearing potential must meet one of the following:

  * Documented postmenopausal (defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments).
  * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy with last menses >1 year ago (excluding tubal ligation, radiation-induced oophorectomy).
  * Documented amenorrhoeic for 12 months (defined as women under the age of 50 years with serum follicle-stimulating hormone (FSH), luteinizing hormone (LH) and plasma oestradiol levels in the postmenopausal range for the institution).
* Patient is willing and able to comply with the protocol for the duration of the trial.

Exclusion Criteria:

* Diagnosis of ataxia-telangiectasia syndrome.
* Women who are pregnant or breast-feeding.
* Women of child-bearing potential and male participants who are unwilling to use 2 highly effective forms of contraception during the trial and for 6 months after the completion of the trial treatment.
* Cytotoxic chemotherapy within 21 days prior to start of trial treatment (greater than 5 half-lives is allowed for washout in patients treated with non-cytotoxic drugs).
* Exposure to a small molecule IMP within 30 days or 5 half-lives (whichever is longer) prior to the start of treatment.
* Palliative radiotherapy within 21 days prior to start of trial treatment.
* Immunotherapy within 42 days prior to start of trial treatment.
* New treatment with bisphosphonates or denosumab for bone metastases within 5 days prior to start of trial treatment (patients can receive a stable dose of bisphosphonates or denosumab for bone metastases before and during the trial as long as these were started at least 5 days prior to start of treatment).
* Major surgery within 2 weeks prior to start of trial treatment (patients must have recovered from any effects of major surgery).
* Current treatment with steroids (doses of >10mg of prednisone or equivalent) or other immunosuppressive drugs within 14 days prior to start of trial treatment.
* Any other malignancy which has been active or treated within the past three years (with the exception of cervical intra-epithelial neoplasia, non-melanoma skin cancer, ductal carcinoma in situ, stage 1 grade 1 endometrial carcinoma, or other solid tumours curatively treated with no evidence of disease for ≥5 years prior).
* Current treatments with known potent cytochrome P (CYP) 3A inhibitors, potent CYP3A inducers, CYP3A4 and/or CYP2B6 substrates with a narrow therapeutic index or Pgp modulators (wash out period of 5 half-lives, but three weeks for St. John's Wort, see Appendix 4). The use of herbal supplements, homeopathic remedies or 'folk remedies' is not permitted.
* Impaired hepatic or renal function defined as:

  * AST or ALT >2.5 x ULN (or 5 times if liver metastasis).
  * Total bilirubin >1.5 x ULN.
  * Glomerular filtration rate (GFR) (calculated by Cockcroft-Gault) of <41 ml/min.
* Inadequate bone marrow reserve or organ function defined as:

  * Absolute neutrophil count <1.5 x 109/L.
  * Platelet count <100 x 109/L with no blood transfusions in the past 28 days.
  * Haemoglobin <90 g/L with no platelet transfusions in the past 28 days.
* INR ≥1.25 above the normal range.
* Haematuria +++.
* Known history of cardiac dysfunction within the last 6 months defined as:

  * Myocardial infarction
  * NYHA Class II/III/IV heart failure
  * Unstable angina pectoris
  * Unstable cardiac arrhythmias not controlled with a pacemaker or medication (e.g. complete left bundle branch block or third degree heart block).
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc) >470 msec for women, and >450 msec for men obtained from 3 electrocardiograms (ECGs) 2-5 minutes apart using the Fridericia formula.
  * Patients with relative hypotension (<90/60 mm Hg) or clinically relevant orthostatic hypotension, including a fall in blood pressure of > 20 mmHg.
  * Patients at risk of brain perfusion problems (e.g. medical history of carotid stenosis, pre-syncope, syncope episodes or a history of transient ischaemic attack).
  * Uncontrolled hypertension (grade 2 or above) requiring clinical intervention.
* Patients unable to swallow orally administered medication and with gastrointestinal disorders likely to interfere with absorption of AZD6738.
* Any other concurrent severe and/or uncontrolled medical condition that places the patient at unacceptable risk of toxicity or non-compliance (examples include, but are not limited to, active bleeding diatheses, renal transplant, uncontrolled major seizure disorder, severe COPD, superior vena cava syndrome, extensive bilateral lung disease on high resolution CT scan, severe Parkinson's disease, active inflammatory bowel disease, psychiatric condition, or active infection (including any patient known to have hepatitis B, hepatitis C, human immunodeficiency virus (HIV) or requiring systemic antibiotics, antifungals or antiviral drugs)). Screening for chronic conditions is not required.
* Prior exposure to an ATR inhibitor.
* A known hypersensitivity to AZD6738 or gemcitabine (e.g. excessive myelosuppression), any excipient of the products, or any contraindication to the combination of anti-cancer agents.
* Any unresolved toxicities from prior therapy of CTCAE grade >1 (with the exception of alopecia and CTCAE grade 2 neuropathy).
* Spinal cord compression (unless asymptomatic, stable, and not requiring steroids for at least 4 weeks prior to start of treatment).
* Brain metastases (unless disease outside the central nervous system (CNS) is present, no clinical evidence of progression since completion of CNS-directed therapy, at least 3 weeks between completion of radiotherapy and start of trial treatment, recovery from significant (Grade ≥ 3) acute toxicity) with no on-going requirement for >10 mg of prednisone per day or an equivalent dose of other corticosteroid. If on corticosteroids, the patient should be receiving a stable dose of corticosteroids started at least 4 weeks prior to treatment).
* Judgment by the Investigator that the patient should not participate in the trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity for the combination of AZD6738 and gemcitabine. | Through study completion
  Number of participants with drug related toxicities reported during Cycle 1 (each cycle is 28 days).

SECONDARY OUTCOMES:
Evaluate anti-tumour effect | Through study completion for an average of 6 months
  CT scan tumour measurement assessments from start of treatment until progression

CONTACTS AND LOCATIONS:
Overall Officials: Duncan Jodrell, Principal Investigator — CRUK Cambridge Institute, University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No